CLINICAL TRIAL: NCT06328478
Title: Predictors of Acute Kidney Injury in Critically Ill Children Admitted to Pediatrics Intensive Care Unit At Assiut University Children Hospital.
Brief Title: Predictors of Acute Kidney Injury in Critically Ill Children Admitted to PICU.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Adel Labib Attia, Resident physician, Assiut University
Other Study IDs: Predictors of AKI in PICU.
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Observational prospective study. — Observational prospective study

SUMMARY:
Predictors of Acute Kidney Injury in critically ill children admitted to PICU during one year.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is defined by a sudden loss of excretory kidney function. AKI is part of a range of conditions summarized as acute kidney diseases and disorders (AKD), in which slow deterioration of kidney function or persistent kidney dysfunction is associated with an irreversible loss of kidney cells and nephrons, which can lead to chronic kidney disease (CKD).

AKI is determined by increased serum creatinine levels >0.3 mg/dl (a marker of kidney excretory function) and reduced urinary output <0.5 ml/Kg for more than 8 h (a quantitative marker of urine production) and is limited to a duration of 7 days and when lasts for >3 months is referred to as chronic kidney disease (CKD). Acute kidney injury (AKI) is associated with poor outcome in critically ill children. The reported incidence rate of AKI in children admitted to pediatric intensive care units (PICUs) ranges from 8% and 89% worldwide. Stage 1 was identified in 24.24% of the AKI cases, stage 2 in 31.03% and stage 3 in 44.71%. The most prevalent cause of AKI was represented by prerenal AKI in 85.64% of the cases, followed by 12.16% renal causes respectively 2.18% postrenal causes. Symptoms of an AKI come on suddenly, over the course of hours or days. They depend on the underlying cause, but some of the most common symptoms include hematuria, fever, rash, bloody diarrhea, severe vomiting, abdominal pain, no urine output or high urine output, pale skin. oedema, puffy eyes and detectable abdominal mass. There are many predisposing factors that lead to AKI for such as gastroenteritis, presence of infection, sepsis, shock, cardiac disease, mechanical ventilation hypoxia and coagulopathy are important predictors for AKI.

Despite significant developments in the management of AKI, the overall mortality rate of patients with AKI has not improved dramatically. The most widely available studies deal primarily with AKI, reporting mortality rates between 11% and 63% in pediatric patients.

Outcomes among children who develop acute kidney injury (AKI). Children who develop AKI while hospitalized are at risk for poorer short- and mid/long-term outcomes. Across both acute and critical care populations, AKI is associated with longer lengths of stay, non-recovery of baseline renal function, and chronic renal disease including proteinuria, hypertension, and chronic kidney disease (CKD)

ELIGIBILITY:
Inclusion Criteria:

* children aged from month to 18 years admitted to PICU between April 2024 to May 2025.

Exclusion Criteria:

* Exclusion of children aged below 1 month and older than 18 years.
* chronic kidney disease.
* renal malformations.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All cases of acute kidney injury in pediatrics from 1 month to 18 years incritically ill Patient admitted to PICU Assiut University Children Hospital during one year of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury and survival to discharge from the PICU. | One year from April 2024 to May 2025

REFERENCES:
- [Background] Kellum JA, Romagnani P, Ashuntantang G, Ronco C, Zarbock A, Anders HJ. Acute kidney injury. Nat Rev Dis Primers. 2021 Jul 15;7(1):52. doi: 10.1038/s41572-021-00284-z. PMID 34267223
- [Background] Basu RK, Kaddourah A, Terrell T, Mottes T, Arnold P, Jacobs J, Andringa J, Goldstein SL; Prospective Pediatric AKI Research Group (ppAKI). Assessment of Worldwide Acute Kidney Injury, Renal Angina and Epidemiology in critically ill children (AWARE): study protocol for a prospective observational study. BMC Nephrol. 2015 Feb 26;16:24. doi: 10.1186/s12882-015-0016-6. PMID 25882434
- [Background] Ciccia E, Devarajan P. Pediatric acute kidney injury: prevalence, impact and management challenges. Int J Nephrol Renovasc Dis. 2017 Mar 29;10:77-84. doi: 10.2147/IJNRD.S103785. eCollection 2017. PMID 28435306
- [Background] Naik S, Sharma J, Yengkom R, Kalrao V, Mulay A. Acute kidney injury in critically ill children: Risk factors and outcomes. Indian J Crit Care Med. 2014 Mar;18(3):129-33. doi: 10.4103/0972-5229.128701. PMID 24701061
- [Background] Duzova A, Bakkaloglu A, Kalyoncu M, Poyrazoglu H, Delibas A, Ozkaya O, Peru H, Alpay H, Soylemezoglu O, Gur-Guven A, Bak M, Bircan Z, Cengiz N, Akil I, Ozcakar B, Uncu N, Karabay-Bayazit A, Sonmez F; Turkish Society for Pediatric Nephrology Acute Kidney Injury Study Group. Etiology and outcome of acute kidney injury in children. Pediatr Nephrol. 2010 Aug;25(8):1453-61. doi: 10.1007/s00467-010-1541-y. Epub 2010 May 30. PMID 20512652
- [Background] Cleto-Yamane TL, Gomes CLR, Suassuna JHR, Nogueira PK. Acute Kidney Injury Epidemiology in pediatrics. J Bras Nefrol. 2019 Apr-Jun;41(2):275-283. doi: 10.1590/2175-8239-JBN-2018-0127. Epub 2018 Nov 14. PMID 30465591
- [Background] Uber AM, Sutherland SM. Acute kidney injury in hospitalized children: consequences and outcomes. Pediatr Nephrol. 2020 Feb;35(2):213-220. doi: 10.1007/s00467-018-4128-7. Epub 2018 Nov 1. PMID 30386936